CLINICAL TRIAL: NCT03455946
Title: Testing the Feasibility of the DASH Cloud Intervention Using Amazon Alexa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D0298
Record Dates: First submitted 2017-12-27; First posted 2018-03-07 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Behavior, Health; Diet Modification
Keywords: Digital Health; Amazon Alexa
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): DASH Cloud with Alexa
  Interventions: Behavioral: DASH cloud with Alexa

INTERVENTIONS:
Behavioral: DASH cloud with Alexa — Participants will download and install the Alexa and Nutritionix application ("app") onto their smartphone and study staff will setup the study-specific account to send data to Duke's software system called Prompt. Participants will be instructed to invoke through voice their dietary intake daily for three months using the Nutritionix app through the Amazon Alexa personal assistant. DASH Cloud will access participant's dietary intake data through the Nutritionix application programing interface (API) for three months. Participants' data will automatically be uploaded from the Nutritionix app via the API that links the device with DASH Cloud. DASH Cloud will run an algorithm and send a daily or weekly feedback text message with a score reflecting DASH adherence for the prior days or week's food consumption using a previously validated scoring system.

SUMMARY:
The DASH diet is a proven behavioral strategy to reduce blood pressure, however, national adherence rates are poor. Using digital health tools may help to improve adoption of the DASH diet. Digital health approaches capitalize on the ubiquitous utilization of mobile technologies and have broad dissemination potential. There have been few efforts to test a DASH intervention via digital, and none using voice-activated technologies (e.g, Amazon Alexa). This proposal will enroll up to 20 participants to leverage a commercial diet tracking application, an existing intervention technology platform and the Amazon Echo Dot to test the feasibility of using DASH Cloud, a digital health intervention, with the Amazon Alexa personal assistant.

DETAILED DESCRIPTION:
Digital health approaches are promising intervention channels for improving DASH diet adherence. Almost all Americans own a mobile phone and 97% of mobile phone owners use text messaging. Digital health approaches can capitalize on the ubiquity of mobile technologies and allow investigators to reach affected populations with highly personalized content at low cost. Despite this ubiquity, interventions using text messaging for hypertension self-management primarily rely on reminders for tracking and medication adherence without diet and physical activity behaviors or feedback. As such, they are less effective. Investigators will establish the feasibility of a novel digital health-based approach for disseminating the DASH diet using the Amazon Alexa personal assistant. The data from this pilot feasibility trial will set the foundation for a larger, fully-powered R01 grant to examine whether DASH Cloud using Alexa can improve health outcomes. The primary aim of this proposal is to test the feasibility of the DASH Cloud intervention using Amazon Alexa.

ELIGIBILITY:
Inclusion Criteria:

* Over 21 years old;
* BMI >18.5 kg/m2;
* Current use of a smartphone with an updated operating system
* Data plan
* Willingness to be texted daily or weekly
* Wifi network at home
* An active email account
* Spoken and written English fluency.

Exclusion Criteria:

* CVD event in prior 6 months
* Active malignancy
* Active psychosis or recent psychiatric institutionalization
* Current pregnancy or lactation
* Current participation in a similar trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Intervention feasibility | 3 months
  Utilization of intervention components at 3 months as indicated by the system usability scale

CONTACTS AND LOCATIONS:
Overall Officials: Dori Steinberg, Ph.D, RD, Principal Investigator — Duke University; Gary Bennett, Ph.D, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided